CLINICAL TRIAL: NCT00138827
Title: A Pilot Randomised Comparison of Bicarbonate Based Mouth Care Versus Biotene Based Mouth Care During Radiotherapy
Brief Title: Mouth Care Regimes During Radiotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St George Hospital, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99/65 Graham
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 1998-05

CONDITIONS: Head and Neck Neoplasms
Keywords: Radiotherapy; Mucositis; Xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Xerostomia | interventions — Biotene; Oral Hygiene

INTERVENTIONS:
Drug: Biotene (mouth care)

SUMMARY:
The purpose of this study is to assess whether Biotene oral care products have a benefit in the treatment of xerostomia and mucositis when compared with conventional bicarbonate mouth care regimes.

DETAILED DESCRIPTION:
Grade III and IV mucositis occurs in 30-60% of patients undergoing head and neck irradiation. Where mucositis is severe a patient's ability to swallow may become significantly compromised and nutritional requirements may not be met.

Xerostomia is often an early side effect of treatment. As salivary tissue is very sensitive to radiation there is often a change in saliva early in the treatment.

New products on the market have claimed to alleviate the symptoms of dry mouth and to help the body's natural defenses reduce the harmful oral bacteria. These products contain the important salivary enzymes lactoperoxidase, lysozyme, lactoferrin and glucose oxidase. Biotene products therefore have the potential to reduce microbial populations which result in radiation caries and periodontal disease and in addition provide relief from the discomfort of xerostomia.

Despite the knowledge surrounding xerostomia in the head and neck irradiation population, its treatment has not been well documented and the question of patient comfort is not well addressed.

Comparisons: This study aims to compare the different mouth care regimes and determine the most effective treatment alternatives during radiotherapy. Patients will be randomised to either Biotene or Bicarbonate-based mouth care regimes. Patients will be stratified according to whether they are receiving radiotherapy alone or chemo irradiation to ensure equal distribution across the different mouth care regimes.

ELIGIBILITY:
Inclusion Criteria:

* Are undergoing oral or pharyngeal irradiation with a cumulative dose > 35Gy with at least 1/2 of the salivary tissue contained within the field of treatment.
* May or may not have undergone surgery.
* Are available for follow-up questionnaires.
* Are English speaking or have an easily accessible interpreter.

Exclusion Criteria:

* No co-morbidities which may result in dry mouth, for example Sjögren syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-11; Study Completion 2003-03

PRIMARY OUTCOMES:
Mid treatment, 2 and 6 weeks post treatment relative to baseline: Oral comfort - dichotomised as difficulty yes/no based on 3 questions
Mucositis - dichotomised
Xerostomia - dichotomised
Pain medications - dichotomised

SECONDARY OUTCOMES:
Oral flora
Oral pH
Salivary flow

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Peter H Graham, Principal Investigator — St George Hospital, Sydney, Australia
Locations (1):
- St George Hospital, Cancer Care Centre, Sydney, New South Wales, Australia